CLINICAL TRIAL: NCT03270488
Title: Effects of Laser Therapy on Pain Intensity for Carpometacarpal Joint Osteoarthritis as a Isolated Treatment. A Randomized (Double-blind) Controlled Trial
Brief Title: Laser Therapy, Pain and Carpometacarpal Joint Osteoarthritis Treatment
Acronym: Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMalaga2
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Thumb Osteoarthritis; Pain; Physical Disorder
Keywords: Thumb; Osteoarthritis; Physical Therapy; Pain
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental): Laser application three times a week for 4 weeks.
  Interventions: Other: Laser
- Placebo group (Placebo Comparator): The same equipment was used with a pen that emits a red guide light and a warning sound, but without the emission of a laser beam.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Laser — Laser (power of 3.0w).
  Arms: Laser Group
Other: Placebo — Laser (power 0,0w)
  Arms: Placebo group

SUMMARY:
Osteoarthritis (OA) is a chronic and prevalent joint disorder with great impact on quality of life and high economic burden. Although a number of conservative therapies have proven to be effective for the management of hand OA, only modest treatment effects were reported for most individual interventions. The aim of the proposed study is to assess the effect of laser therapy on pain, function and force in patients with carpometacarpal osteoarthritis (CMC OA).

DETAILED DESCRIPTION:
A randomized, controlled, single-center, double-blind, clinical trial, with 1:1 allocation ratio, were carried out involving patients diagnosis of CMC joint OA grade 1-2 (aged 18 years and above). Both assessor and statistician remained blinded. The research diagnostic criteria for carpometacarpal joint osteoarthritis was used to assess all individuals who agree to participate. All participants were submitted to a clinical examination and X-ray assessment of thumb base to determine carpometacarpal osteoarthritis grade. Based on the clinical and radiological findings, the participants were classified by a rheumatology. Those with CMC OA grade 2-3 were included in the study. The experimental group received laser therapy and control group received a placebo treatment.

The primary outcome measures was pain scores during daily living activities (DLA)- at the base of the thumb measured with VAS (Unidimensional measure of pain: 0-10 (0, no pain and 10, worst pain), and changes in hand function measured using the Quick-Dash questionnaire. Secondary outcome measures included changes in pinch strength. All outcome measures were collected at baseline, immediately following the intervention at 4 weeks and at 12 weeks following the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 diagnosis of CMC joint OA in their dominan hand.
* State 1-2 according to the American College of Rheumatology.
* Pain intensity during activities of daily living (ADLs) of up to 4 of 10 on the visual analog scale (VAS)
* Ability to read or understand the patient information sheets.
* Ability to sign a consent form will be included in the study

Exclusion Criteria:

* Neurologic disorder affecting the upper limb
* Previous treatment for their hand problem in the last 6 months including an intra-articular joint injection to wrist, fingers, or thumb
* Had fractures or a significant hand injury or previous surgery to the wrist, thumb or hand
* Finger tenosynovitis.
* Dupuytren disease.
* Psychological treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 months
  VAS has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' and the right-hand anchor reads 'worst possible pain'; the patients marked a line to represent their pain level. EVA scale was development by Huskisson in 1974. Ensen MP, Karoly P. Self-report scales and procedures for assessing pain in adults. In: Turk DC, Melzack R (eds). Handbook of Pain Assessment. 2nd ed. New York, NY: The Guilford Press, 2001. pp. 15-34.
  Seymour RA. The use of pain scales in assessing the efficacy ofanalgesics in post-operative dental pain. Eur J Clin Pharmacol. 1982;23:441-4 Gatson-Johansson F. Measurement of pain: the psychometric properties of the Pain-O-Meter, a simple, inexpensive pain assessment tool that could change health care practices. J Pain Symptom Manage. 1996;12:172-81.

SECONDARY OUTCOMES:
Key pinch strength | 3 months
  For measure pinch key we used Key pinch dynamometer. Pinch strength was less in patients with early thumb CMC OA. Key pinch had the most robust association with OA diagnosis. Tomas J et al. Weaker Functional Pinch Strength Is Associated With Early Thumb Carpometacarpal Osteoarthritis. Clin Orthop Relat Res (2016) 474:557-561 MacDermid JC, Wessel J, MacIntyre N, Galea V. The relationship between impairment, dexterity and self-reported disability of persons with osteoarthritis of the hand. J Hand Ther. 2008;21:427-8

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Cantero, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cantero-Tellez R, Villafane JH, Valdes K, Garcia-Orza S, Bishop MD, Medina-Porqueres I. Effects of High-Intensity Laser Therapy on Pain Sensitivity and Motor Performance in Patients with Thumb Carpometacarpal Joint Osteoarthritis: A Randomized Controlled Trial. Pain Med. 2020 Oct 1;21(10):2357-2365. doi: 10.1093/pm/pnz297. PMID 31807782